CLINICAL TRIAL: NCT04130282
Title: A Phase Ia Study to Assess Safety and Immunogenicity of the Plasmodium Falciparum Malaria Vaccine Candidate Pfs25-IMX313 in Matrix-M1 Adjuvant in Healthy Adults Living in the UK
Brief Title: VAC077: Safety and Immunogenicity of the Pfs25-IMX313/Matrix-M Vaccine
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Delays caused by Covid-19
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VAC077
Record Dates: First submitted 2019-10-08; First posted 2019-10-17 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Malaria,Falciparum
Keywords: Pfs25
MeSH Terms: conditions — Malaria, Falciparum | interventions — Matrix-M

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group 1 (Experimental): 8 volunteers receiving 3 doses of 10µg Pfs25-IMX313 in 50 µg Matrix-M1 on days 0, 28 and 56
  Interventions: Biological: Pfs25-IMX313/Matrix-M1

INTERVENTIONS:
Biological: Pfs25-IMX313/Matrix-M1 — 3 doses of 10µg Pfs25-IMX313 in 50 µg Matrix-M1 on days 0, 28 and 56

SUMMARY:
This is an open label, single-site, first-in-human, Phase Ia study to assess safety and immunogenicity of the Plasmodium falciparum malaria vaccine candidate Pfs25-IMX313 in Matrix-M1 adjuvant in healthy adults living in the UK

Volunteers will receive 3 doses of vaccine over 2 months and will be followed up for approximately 8 months.

DETAILED DESCRIPTION:
This Phase 1a clinical trial is designed primarily to assess the safety and tolerability of the Pfs25-IMX313/Matrix-M transmission blocking vaccine in healthy adult volunteers. An important secondary objective is to to assess the immune response to the vaccine.

8 volunteers will receive 3 doses of 10µg Pfs25-IMX313 in 50 µg Matrix-M1 on days 0, 28 and 56. Blood samples will be taken for safety testing and to collect information about the immune response. Any symptoms that occur after vaccination will also be recorded.

Healthy volunteers aged 18-45 will be recruited in England at the Centre for Clinical Vaccinology and Tropical Medicine, Churchill Hospital, Oxford.

ELIGIBILITY:
Inclusion Criteria:

The volunteer must satisfy all the following criteria to be eligible for the study:

* Healthy adult aged 18 to 45 years.
* Able and willing (in the Investigator's opinion) to comply with all study requirements.
* Willing to allow the Investigators to discuss the volunteer's medical history with their General Practitioner.
* Women only: Must practice continuous effective contraception for the duration of the study
* Agreement to refrain from blood donation for the duration of the study
* Written informed consent to participate in the trial.

Exclusion Criteria:

The volunteer may not enter the study if any of the following apply:

* History of clinical malaria (any species).
* Travel to a clearly malaria endemic locality during the study period or within the preceding six months.
* Use of immunoglobulins or blood products (e.g., blood transfusion) at any time in the past.
* Receipt of any vaccine in the 30 days preceding enrolment, or planned receipt of any other vaccine within 30 days following each vaccination
* Receipt of an investigational product in the 30 days preceding enrolment, or planned receipt during the study period.
* Concurrent involvement in another clinical trial or planned involvement during the study period
* Prior receipt of an investigational vaccine likely to impact on interpretation of the trial data, as assessed by the Investigator
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed).
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine (e.g. egg products)
* Any history of anaphylaxis in reaction to vaccinations
* Pregnancy, lactation or intention to become pregnant during the study.
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
* History of serious psychiatric condition that may affect participation in the study.
* Any other serious chronic illness requiring hospital specialist supervision.
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 25 standard UK units every week.
* Suspected or known injecting drug abuse in the 5 years preceding enrolment.
* Hepatitis B surface antigen (HBsAg) detected in serum.
* Seropositive for hepatitis C virus (antibodies to HCV) at screening or (unless has taken part in a prior hepatitis C vaccine study with confirmed negative HCV antibodies prior to participation in that study, and negative HCV RNA PCR at screening for this study).
* Volunteers unable to be closely followed for social, geographic or psychological reasons.
* Any clinically significant abnormal finding on biochemistry or haematology blood tests, urinalysis or clinical examination.
* Any other significant disease, disorder, or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.
* Inability of the study team to contact the volunteer's GP to confirm medical history and safety to participate.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
Assessment of safety and reactogenicity through collection of data on the frequency, duration and severity of solicited and unsolicited adverse events. | 8 months
  The following parameters will be assessed:
  * Frequency, duration and severity of solicited local reactogenicity signs and symptoms for 7 days following each vaccination
  * Frequency, duration and severity of solicited systemic reactogenicity signs and symptoms for 7 days following the vaccination
  * Frequency, duration and severity of unsolicited adverse events for 28 days following the vaccination
  * Change from baseline for safety haematological and biochemical laboratory measures, which will presented according to local grading scales, for 28 days following vaccination
  * Frequency, duration and severity of serious adverse events during the whole study duration

SECONDARY OUTCOMES:
Humoral and cellular immunogenicity of the Pfs25-IMX313/Matrix-M1 vaccine, when administered to healthy adult volunteers | 8 months
  Pfs25-specific immunogenicity will be assessed by immunological assays, with comparison before and after vaccination. The main outcome measures will be humoral and B cell responses to the Pfs25 protein - total IgG, isotypes and avidity; T cell responses to Pfs25 by ex vivo ELISpot and flow cytometry assays.
Ex-vivo efficacy of the Pfs25-IMX313/Matrix-M1 vaccine, when administered to healthy adult volunteers | 8 months
  Ex vivo functional blocking activity of purified IgG against the P. falciparum NF54 strain will be assessed by standard membrane feeding assay.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Minassian, PhD, Principal Investigator — University of Oxford
Locations (1):
- CCVTM, University of Oxford, Churchill Hospital, Oxford, United Kingdom